CLINICAL TRIAL: NCT00541866
Title: Phase 1b/2, Open-Label, Multicenter, Dose-Escalating, Clinical Study of the Safety, Tolerability, and PK and PD Profiles of Voreloxin Injection in Combination With Cytarabine in Patients With Relapsed or Refractory AML
Brief Title: Safety and Tolerability Study of Voreloxin and Cytarabine Combination in Acute Myeloid Leukemia in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0012
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Acute Myeloid; Relapsed; Refractory; Cancer; AML; Cytarabine; SNS-595; Phase 1; Voreloxin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence; Neoplasms | interventions — vosaroxin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voreloxin injection and cytarabine (Experimental): Dose-escalation Phase
  * Schedule A:
  * Schedule B:
  Expansion Phase
  * Schedule A:
  * Schedule B:
  Interventions: Drug: Voreloxin injection and cytarabine

INTERVENTIONS:
Drug: Voreloxin injection and cytarabine — Dose-escalation Phase
  * Schedule A: vosaroxin injection (dose-escalation from 10 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (24-hour CIV infusion of 400 mg/m2/day × 5 days)
  * Schedule B: vosaroxin injection (dose-escalation from 70 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days)
  Expansion Phase The MTD determined in the dose-escalation phase was used in the expansion phase.
  * Schedule A: 80 mg/m2 vosaroxin on Days 1 and 4 in combination with cytarabine (24-hour CIV infusion at 400 mg/m2/day × 5 days)
  * Schedule B: 90 mg/m2 vosaroxin (dose-escalation) on Days 1 and 4 in combination with cytarabine (2 hour IV infusion at 1 g/m2/day × 5 days)
  Other Names: ARA-C, Cytosar-U

SUMMARY:
This study will evaluate the safety and tolerability of voreloxin (vosaroxin) injection in combination with cytarabine in patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
An open-label, Phase 1b/2 study using a dose-escalation design with expansion at the maximum tolerated dose (MTD) using 2 dosing schedules:

During the Schedule A dose-escalation phase, patients with relapsed or refractory acute myeloid leukemia (AML) enrolled in cohorts of at least 3 patients to identify the MTD. Begin with a starting dosing regimen of vosaroxin of 10 mg/m2 on Days 1 and 4 of each cycle in combination with a 24-hour continuous intravenous (CIV) infusion of cytarabine 400 mg/m2/day × 5 days. If none of the 3 patients or 1 of 6 patients experience a dose-limiting toxicity (DLT) at the vosaroxin starting dose, dose-escalate vosaroxin. If 2 of 6 patients experienced a DLT at the vosaroxin starting dose, reduce the dose of cytarabine to reduced to 200 mg/m2 (only case in which the cytarabine could have been reduced). The vosaroxin dose escalated following a modified Fibonacci schema.

For Schedule B dose-escalation phase, patients with relapsed or refractory AML enrolled in cohorts of at least 3 patients to identify the MTD. Begin with a starting dose regimen of vosaroxin of 70 mg/m2 on Days 1 and 4 in combination with cytarabine as a 2-hour infusion of 1 g/m2/day × 5 days. No reductions of cytarabine allowed in Schedule B. If none of the 3 patients or 1 of 6 patients experienced a DLT in the first cohort of Schedule B, escalate the dose of vosaroxin. If DLTs occurred in 2 of 6 patients during the starting dose, reduce the vosaroxin dose to 50 mg/m2.

For both Schedules, the highest dose at which fewer than 2 of 6 patients experienced a DLT during induction became the MTD and the recommended future dose.

Once the MTD of vosaroxin was determined for Schedule A, first relapse patients were enrolled in the expansion phase at that dose level to obtain additional safety and efficacy information. When the MTD of vosaroxin was determined for Schedule B, first relapse patients and patients with primary refractory disease were enrolled in the expansion phase at that dose level to characterize the safety and efficacy profile in this population.

ELIGIBILITY:
KEY INCLUSION CRITERIA

1. Relapsed or refractory AML subtypes defined by WHO, except acute promyelocytic leukemia. Relapsed/refractory disease may be de novo AML or secondary AML
2. Treated with one to threee induction/reinduction AML regimens, prior induction or consolidation therapy with cytarabine allowed
3. At least 10% blasts by BM biopsy or aspirate
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
5. Clinical laboratory values of a) Serum creatinine ≤1.5 mg/dL and calculated or measured creatinine clearance (CRcl) of ≥50 mL/min, b) Total bilirubin ≤1.5 X upper limit of normal and c) Aspartate aminotransferase (AST) or alkaline phosphatase ≤2.5 X ULN.

KEY EXCLUSION CRITERIA

Patients with:

1. Allogenic bone marrow transplant/stem cell transplant
2. Persistent, clinically significant, chronic toxicities from prior AML therapy that would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with study procedures
3. Acute promyelocytic leukemia
4. Disseminated intravascular coagulation
5. Active infections, unless adequately treated with antibiotic, antiviral, or antifungal agents within in 7 days before Induction Day 1
6. Active central nervous system involvement by AML
7. Other active malignancies or other malignancies within the last 12 months except nonmelanoma skin cancer or cervical intraepithelial neoplasia
8. A requirement for hemodialysis or peritoneal dialysis
9. A history of myocardial infarction within the 3 months before treatment with vosaroxin
10. A history of cerebrovascular accident/transient ischemic attack within the 3 months before treatment with vosaroxin
11. A thromboembolic event (deep vein thrombosis or pulmonary embolus) within 28 days before treatment with vosaroxin
12. Investigational products taken within 28 days before treatment with vosaroxin, and non-investigational cancer therapies or radiation therapy within 14 days before treatment with vosaroxin, with the exception of hydroxyurea.
13. A known intolerance to cytarabine or known allergy to D-sorbitol or methanesulfonic acid (excipients used in vosaroxin)
14. Prior exposure to vosaroxin
15. Any other medical, psychological, or social condition that contraindicates their participation in the clinical study due to safety concerns or compliance with study procedures in the opinion of the Investigator,or Sunesis Medical Monitor

    In addition:
16. Women who are pregnant or breastfeeding
17. Women who are of childbearing potential or male patients who had partners of childbearing potential who were unwilling to use an approved, effective means of contraception according to the study site's standards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-10-06 (Actual); Primary Completion 2012-02-15 (Actual); Study Completion 2012-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunesis Medical Monitor, MD, Study Director — Sunesis Pharmaceuticals
Locations (9):
- United States (9):
  - HealthOne Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University - Sidney Kimmel Cancer Center, Baltimore, Maryland
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Aggregate data of Adverse Events

REFERENCES:
- [Derived] Lancet JE, Roboz GJ, Cripe LD, Michelson GC, Fox JA, Leavitt RD, Chen T, Hawtin R, Craig AR, Ravandi F, Maris MB, Stuart RK, Karp JE. A phase 1b/2 study of vosaroxin in combination with cytarabine in patients with relapsed or refractory acute myeloid leukemia. Haematologica. 2015 Feb;100(2):231-7. doi: 10.3324/haematol.2014.114769. Epub 2014 Nov 7. PMID 25381131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted in 7 centers in the USA between 2007 and 2010
Pre-assignment Details: Dose-escalation phase Group 1 (Sch A, 10 to 90 mg/m2): 41 patients (39 treated) Group 2 (Sch B, 70 to 90 mg/m2): 18 patients
  Dose-expansion phase Group 3 (Sch A first relapse, 80 mg/m2): 17 patients Group 4 (Sch B first relapse, 90 mg/m2): 16 patients Group 5 (Sch B primary refractory, 90 mg/m2): 18 patients Total: 110. Treated: 108
Groups:
- Group 1 (Sch A, 10 to 90 mg/m2): Dose Escalation Phase Schedule A: vosaroxin injection (dose-escalation from 10 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Group 2 (Sch B, 70 to 90 mg/m2):: Dose Escalation Phase Schedule B: vosaroxin injection (dose-escalation from 70 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days)
- Group 3 (Sch A, First Relapse, 80 mg/m2): Expansion Phase: Schedule A: 80 mg/m2 vosaroxin on Days 1 and 4 in combination with cytarabine (24-hour CIV infusion at 400 mg/m2/day × 5 days)
- Group 4 (Sch B, First Relapse, 90 mg/m2): Expansion Phase: Schedule B: 90 mg/m2 vosaroxin (dose-escalation) on Days 1 and 4 in combination with cytarabine (2 hour IV infusion at 1 g/m2/day × 5 days)
- Group 5 (Sch B, Primary Refractory, 90 mg/m2): Expansion Phase Schedule B: 90 mg/m2 vosaroxin (dose-escalation) on Days 1 and 4 in combination with cytarabine (2 hour IV infusion at 1 g/m2/day × 5 days)
Period: Overall Study
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2) | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2)
Started | 41 (41 started, but only 39 treated) | 18 | 17 | 16 | 18
Completed | 7 | 0 | 2 | 0 | 3
Not Completed | 34 | 18 | 15 | 16 | 15
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 19 | 15 | 10 | 12 | 14
Not completed — Not Reported or Other | 11 | 3 | 3 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Sch A, 10 to 90 mg/m2); Group 3 (Sch A, First Relapse, 80 mg/m2):: Schedule A: vosaroxin injection (dose-escalation from 10 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Group 2 (Sch B, 70 to 90 mg/m2):; Group 4 (Sch B, First Relapse, 90 mg/m2); Group 5 (Sch B, Primary Refractory, 90 mg/m2):: Schedule B: vosaroxin injection (dose-escalation from 70 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days)
- Total: Total of all reporting groups
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2): | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2): | Total
Number analyzed (Participants) | 39 | 18 | 17 | 16 | 18 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (10.90) | 47.4 (13.83) | 59.7 (9.29) | 58.4 (11.03) | 56.3 (12.09) | 56.3 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 6 | 6 | 8 | 36
  Male | 28 | 13 | 11 | 10 | 10 | 72
Region of Enrollment [Number; unit: participants]
  United States | 39 | 18 | 17 | 16 | 18 | 108

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-Limiting Toxicity (DLT) to Determine Maximum Tolerated Dose in Schedule A and Schedule B of Dose Escalation Phase (Group 1 and Group 2)
Description: Patients were treated in cohorts with escalating doses of vosaroxin administered in combination with cytarabine in Schedule A, and with vosaroxin in escalating doses in Schedule B. For both Schedules, the highest dose at which fewer than 2 of 6 (<0.33) patients experienced a dose-limiting toxicity (DLT) during induction became the MTD and the recommended future dose.
Time Frame: From start of treatment (Day 1) through Induction Day 29 or the start of reinduction, whichever occurred first.
Population: Patients experiencing a dose-limiting toxicity (DLT) during induction when treated with escalating doses of vosaroxin administered in combination with cytarabine on Days 1 and 4 in Schedule A, and with vosaroxin in escalating doses administered on Days 1 and 4 in Schedule B.
Measure: Count of Participants; unit: Participants
Groups:
- Sch A, Cohort 10mg/m2: Vosaroxin injection 10 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch A, Cohort 20mg/m2: Vosaroxin injection 20 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- SchA, Cohort 34mg/m2: Vosaroxin injection 34 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch A, Cohort 50mg/m2: Vosaroxin injection 50 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch A, Cohort 70mg/m2: Vosaroxin injection 70 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch A, Cohort 80mg/m2; Sch B, Cohort 80mg/m2: Vosaroxin injection 80 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch A, Cohort 90mg/m2; Sch B, Cohort 90mg/m2: Vosaroxin injection 90 mg/m2 on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Sch B, Cohort 70 mg/m2: Schedule B: vosaroxin injection 70 mg/m2 on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days).
Arm/Group | Sch A, Cohort 10mg/m2 | Sch A, Cohort 20mg/m2 | SchA, Cohort 34mg/m2 | Sch A, Cohort 50mg/m2 | Sch A, Cohort 70mg/m2 | Sch A, Cohort 80mg/m2 | Sch A, Cohort 90mg/m2 | Sch B, Cohort 70 mg/m2 | Sch B, Cohort 80mg/m2 | Sch B, Cohort 90mg/m2
Number analyzed (Participants) | 4 | 3 | 4 | 6 | 7 | 8 | 7 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1

2. Secondary Outcome: Remission Rates (CR+CRp)
Description: Complete remission (CR) plus CR with incomplete platelet recovery (CRp) per The IWG criteria for remission modified by Sunesis, assessed by investigator.
  CR is defined as >1000 Neutrophils (ul), >100,000 Platelets (uL) and <5 BM Blasts (%); CRp is defined as >1000 Neutrophils (ul), <=100,000 Platelets (uL) and <5 BM Blasts (%); CRi is defined as >1000 Neutrophils (ul), <100,000 Platelets (uL) and <5 BM Blasts (%); Investigators were to determine a response category for each patient by examination of bone marrow and blood counts at the time of hematologic recovery after induction or reinduction. Investigator assessment categories included CR, CRp, CRi (CR with morphologic CR with incomplete blood count recovery), PR (partial remission), treatment failure, and relapse.
Time Frame: Monthly after the end of treatment for the first year, then every 2 months thereafter for upto 2 years
Population: All treated set which includes all enrolled patients who received any IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Total: 5 groups combined
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2): | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2): | Total
Number analyzed (Participants) | 39 | 18 | 17 | 16 | 18 | 108
Participants | 9 | 4 | 7 | 3 | 4 | 27

3. Secondary Outcome: Leukemia-free Survival (LFS)
Description: Leukemia-free survival is censored at the last known alive date without report of relapse.
Time Frame: From time of the start of CR or CRp to the earliest date of relapse, commencement of reinduction therapy, or death, assessed monthly up to 2 years after the end of study visit.
Population: All treated analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2): | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2):
Number analyzed (Participants) | 39 | 18 | 17 | 16 | 18
months | 12.0 [4.0 to 32.7] | 4.7 [2.3 to 25.2] | 7.4 [0.5 to 25.6] | 25.2 [2.1 to 26.6] | NA [9.3 to NA] — The median and upper confidence Interval were not available due to insufficient number of participants with events

4. Secondary Outcome: Overall Survival
Description: Overall survival is censored at the earlier of the cutoff date for analysis and the last date known to be alive for patients not known to have died.
Time Frame: Time between the date of first study treatment and the date of death due to any cause for upto 2 years after the end of study visit
Population: All treated analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2): | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2):
Number analyzed (Participants) | 39 | 18 | 17 | 16 | 18
months | 4.1 [2.5 to 8.5] | 8.0 [3.3 to 13.3] | 4.1 [2.5 to 11.8] | 7.1 [4.3 to 13.6] | 5.9 [2.9 to 16.4]

5. Secondary Outcome: All Cause Mortality
Description: Mortality of those patients enrolled in the study and receiving intervention
Time Frame: 30 and 60 days
Population: All treated analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2) | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2) | Group 4 (Sch B, First Relapse, 90 mg/m2) | Group 5 (Sch B, Primary Refractory, 90 mg/m2)
Number analyzed (Participants) | 39 | 18 | 17 | 16 | 18
Participants
  30 Days | 8 | 0 | 1 | 0 | 1
  60 Days | 10 | 2 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: 4 years, 4 months
Groups:
- Group 1 (Sch A, 10 to 90 mg/m2):; Group 3 (Sch A, First Relapse, 80 mg/m2): Schedule A: vosaroxin injection (dose-escalation from 10 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (24-hour continuous IV [CIV] infusion of 400 mg/m2/day × 5 days)
- Group 2 (Sch B, 70 to 90 mg/m2):: saroxin injection (dose-escalation from 70 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days)
- Group 4 (Sch B, First Relapse, 90 mg/m2):; Group 5 (Sch B, Primary Refractory, 90 mg/m2):: Schedule B: vosaroxin injection (dose-escalation from 70 to 90 mg/m2) on Days 1 and 4 in combination with cytarabine (2-hour intravenous [IV] infusion of 1 g/m2/day × 5 days)
Arm/Group | Group 1 (Sch A, 10 to 90 mg/m2): | Group 2 (Sch B, 70 to 90 mg/m2): | Group 3 (Sch A, First Relapse, 80 mg/m2) | Group 4 (Sch B, First Relapse, 90 mg/m2): | Group 5 (Sch B, Primary Refractory, 90 mg/m2):
All-Cause Mortality (participants affected / at risk) | 36/39 | 16/18 | 15/17 | 14/16 | 13/18
Serious Adverse Events (participants affected / at risk) | 20/39 | 7/18 | 9/17 | 3/16 | 11/18
Other Adverse Events (participants affected / at risk) | 39/39 | 18/18 | 17/17 | 16/16 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Sch A, 10 to 90 mg/m2): (N=39) | Group 2 (Sch B, 70 to 90 mg/m2): (N=18) | Group 3 (Sch A, First Relapse, 80 mg/m2) (N=17) | Group 4 (Sch B, First Relapse, 90 mg/m2): (N=16) | Group 5 (Sch B, Primary Refractory, 90 mg/m2): (N=18)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 0 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 1 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 2 | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Sch A, 10 to 90 mg/m2): (N=39) | Group 2 (Sch B, 70 to 90 mg/m2): (N=18) | Group 3 (Sch A, First Relapse, 80 mg/m2) (N=17) | Group 4 (Sch B, First Relapse, 90 mg/m2): (N=16) | Group 5 (Sch B, Primary Refractory, 90 mg/m2): (N=18)
Anaemia (Blood and lymphatic system disorders) | 19 | 11 | 8 | 11 | 6
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 12 | 8 | 10 | 8
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 2 | 6 | 5
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 9 | 7 | 9 | 8
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 7 | 0 | 2 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Intracardiac mass (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 2 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 11 | 6 | 4 | 3 | 6
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Auricular swelling (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 5 | 0 | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1
Mastoid disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 2 | 2 | 2 | 3
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 1 | 0
Eye irritation (Eye disorders) | 2 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 1
Meibomianitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 1 | 1 | 0
Ocular icterus (Eye disorders) | 2 | 0 | 0 | 0 | 1
Orbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 2 | 0 | 0 | 0 | 0
Pupil fixed (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 11 | 2 | 4 | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 15 | 4 | 4 | 1 | 8
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0
Anal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 8 | 8 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 28 | 13 | 15 | 12 | 12
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 4 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 6 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces hard (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 5 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 29 | 6 | 14 | 10 | 12
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 1
Oral mucosal petechiae (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Oral soft tissue disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 4 | 4 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 21 | 13 | 11 | 15 | 10
Tongue coated (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 21 | 7 | 11 | 4 | 9
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Application site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0
Application site vesicles (General disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 11 | 3 | 8 | 1 | 8
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0
Catheter related complication (General disorders) | 1 | 4 | 2 | 5 | 2
Catheter site erythema (General disorders) | 4 | 2 | 2 | 2 | 0
Catheter site excoriation (General disorders) | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 3 | 2 | 0 | 1 | 1
Catheter site oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 4 | 2 | 2 | 0 | 1
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 1 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 3 | 1 | 1 | 1 | 0
Chest pain (General disorders) | 4 | 1 | 1 | 0 | 2
Chills (General disorders) | 18 | 8 | 8 | 6 | 7
Face oedema (General disorders) | 4 | 1 | 0 | 0 | 2
Facial pain (General disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 16 | 7 | 7 | 3 | 9
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 2 | 0 | 1 | 2 | 1
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion site vesicles (General disorders) | 2 | 0 | 0 | 0 | 0
Infusion site warmth (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 3 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0 | 1 | 2
Oedema peripheral (General disorders) | 17 | 3 | 7 | 3 | 9
Pain (General disorders) | 5 | 3 | 4 | 4 | 3
Performance status decreased (General disorders) | 0 | 0 | 2 | 1 | 0
Pyrexia (General disorders) | 13 | 6 | 2 | 1 | 3
Sensation of foreign body (General disorders) | 1 | 0 | 0 | 0 | 0
Suprapubic pain (General disorders) | 1 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0 | 1
Upper extremity mass (General disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 5 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Anorectal cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anorectal infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 3 | 1
Clostridial infection (Infections and infestations) | 3 | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 2 | 0 | 4 | 2 | 1
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 2 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 2 | 3 | 3 | 3 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Torulopsis infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 2 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulval cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Chemical eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 6 | 2 | 2 | 5 | 2
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 1 | 2
Vertebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 0
Bacteria sputum identified (Investigations) | 0 | 0 | 1 | 0 | 0
Bacteria stool identified (Investigations) | 2 | 0 | 1 | 0 | 0
Bacteria urine identified (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 9 | 4 | 2 | 0 | 2
Bronchoscopy abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 2 | 1 | 1 | 0 | 2
Computerised tomogram abdomen abnormal (Investigations) | 2 | 0 | 0 | 0 | 0
Computerised tomogram abnormal (Investigations) | 2 | 1 | 2 | 1 | 0
Culture stool positive (Investigations) | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 0 | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 1 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1 | 0 | 0
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Occult blood (Investigations) | 0 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 1 | 0 | 0
Ultrasound kidney (Investigations) | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 2 | 1
Varicella zoster virus serology positive (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 4 | 2 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 12 | 11 | 13 | 5 | 10
Cachexia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 2 | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 4 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 4 | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 3 | 4 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 10 | 15 | 9 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 10 | 13 | 7 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 0 | 9 | 5 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 4 | 4 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 3 | 2 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 7 | 3 | 4 | 7 | 2
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 5 | 1 | 3 | 1 | 5
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 14 | 7 | 3 | 7 | 5
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 0 | 1 | 0
Hyposmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 1 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 1 | 1 | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 2 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 7 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 11 | 6 | 6 | 5 | 3
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 6 | 1 | 2 | 0 | 4
Delirium (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 6 | 1 | 5 | 1 | 3
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 2 | 1 | 1 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 3 | 1 | 1 | 2 | 1
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 14 | 3 | 9 | 6 | 5
Mental status changes (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 3 | 1 | 1 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 4
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1
Renal failure acute (Renal and urinary disorders) | 4 | 0 | 2 | 2 | 0
Urethral pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 1 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Scrotal irritation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal laceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3 | 4 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 2 | 2 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 4 | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 7 | 4 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 4
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0 | 1 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 3 | 5 | 6 | 3
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 3 | 2 | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 4 | 2 | 0 | 2
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2 | 1 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2 | 1 | 3 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 3 | 7 | 3 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 0
Post procedural drainage (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 6 | 0 | 1 | 2 | 1
Haematoma (Vascular disorders) | 2 | 1 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 8 | 3 | 1 | 3 | 3
Hypotension (Vascular disorders) | 17 | 8 | 7 | 7 | 7
Jugular vein distension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 5 | 1 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Vascular calcification (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vasodilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Further study is needed to confirm the results due to limited sampling size. Statistical fields are not included here because no statistical testings were performed to compare any of the treatment groups. No p-values or odds ratios were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days